CLINICAL TRIAL: NCT07184073
Title: Association Between Cognitive Fraility and Blood and CSF Biomarkers in Older Orthopedic Patients Under Regional Anesthesia
Brief Title: Cognitive Fraility and Biomarkers in Older Patients
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, ELVIN KESIMCI, prof. dr, Baskent University
Other Study IDs: KA21/124
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment; Frail Older Adults; Orthopaedic Surgery
Keywords: cognitive frailty; neurofilament light chain; cerebrospinal fluid biomarkers; older adult patients; orthopedic surgery
MeSH Terms: conditions — Cognitive Dysfunction; Charcot-Marie-Tooth disease, Type 1F | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — samples of cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- age 65-74
  Interventions: Behavioral: assessment Mini mental state examination; Behavioral: assessment FRAIL scale; Other: collecting cerebrospinal fluid during regional anesthesia

INTERVENTIONS:
Behavioral: assessment Mini mental state examination — pre operatively four weeks postoperatively
Behavioral: assessment FRAIL scale — pre operatively four weeks postoperatively
Other: collecting cerebrospinal fluid during regional anesthesia — In the operating room regional anesthesia was administered according to the surgical plan

SUMMARY:
this study aimed to investigate the association between cognitive fraility and selected plasma and cerebrospinal fluid biomarkers related to neurodegenetaion and neuroinflammation in older adult patients undergoing elective orthopedic surgery.

The main questions it aims to answer is:

* Can biomarkers indicating neurodegeneration and neuroinflammation be correlated with preoperative frailty and cognitive functions?
* Can these biomarkers be used as potential tools for early identification in vulnarable populations?

DETAILED DESCRIPTION:
It is a cross sectional study

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients
* >65 age patients

Exclusion Criteria:

* history of psychiatric or neurological disease
* uncontrolled hypertension
* alchohol dependence
* renal failure
* active liver disease
* cancer-related or emergency surgery
* unwillingness to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged 65 years or older who underwent elective major lower extremity orthopedic surgery under regional anesthesia
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
Correlation between biomarkers of neurodegeneration and preoperative frailty, cognitive function? | preoperatively and four weeks postoperatively
  p<0,05 was accepted as statistically significant

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fang J, Liang H, Chen M, Zhao Y, Wei L. Association of preoperative cognitive frailty with postoperative complications in older patients under general anesthesia: a prospective cohort study. BMC Geriatr. 2024 Oct 19;24(1):851. doi: 10.1186/s12877-024-05431-1. PMID 39427111